CLINICAL TRIAL: NCT02544191
Title: GnRHa Combined With hCG and hMG for Treatment of Patients With Non-obstructive Azoospermia: A Single-center Prospective Study in China
Brief Title: GnRHa Combined With hCG and hMG for Treatment of Patients With Non-obstructive Azoospermia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Bing Yao, Director of Center for Reproductive Medicine, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AzoospermiaNanjing
Record Dates: First submitted 2015-08-29; First posted 2015-09-09 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Azoospermia
Keywords: azoospermia nonobstructive; male infertility
MeSH Terms: conditions — Azoospermia; Azoospermia, Nonobstructive; Infertility, Male | interventions — Goserelin; Chorionic Gonadotropin; Urofollitropin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GnRHa/ hCG/ hMG (Experimental): 3.6mg GnRHa (Goserelin, AstraZeneca UK Limited) every 28days for 5 months. After 2 months from the first Goserelin injection, all subjects were treated with hCG (Pregnyl, N.V. Organon Oss,Holland ) at a dose of 2000 IU once a week for 3 months. After 3 months from the first Goserelin injection, all subjects were treated with hMG (Urofollitropin for Injection, Livzon Pharm Group Inc., China) at a dose of 150 IU every 3 days for 2 months.
  Interventions: Drug: GnRHa/ hCG/ hMG

INTERVENTIONS:
Drug: GnRHa/ hCG/ hMG — GnRHa was injected subcutaneously at a dose of 3.6mg every 28 days for 5 months. After 2 months from the first GnRHa injection, all subjects were treated with hCG at a dose of 2000 IU once a week for 3 months. After 3 months from the first Goserelin injection, all subjects were treated with hMG at a dose of 150 IU every 3 days for 2 months.
  Other Names: Goserelin/ Pregnyl/ Urofollitropin for Injection

SUMMARY:
Preliminary reports showed that hormonal treatment may improve the chance of retrieving viable testicular sperm from men with NOA. It was generally believed that gonadotrophin treatment would be ineffective in the presence of high plasma levels of endogenous gonadotrophin.The purpose of this study is to determine whether GnRHa(gonadotropin-releasing hormone agonist) combined with hCG(human chorionic gonadotropin) and hMG(human menopausal gonadotropin) are effective in the treatment of non-obstructive azoospermia.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-45 with clinical diagnosis of non-obstructive azoospermia.
* At least testicular volume more than 8.0ml on one side .
* FSH more than 5.5 IU/L.

Exclusion Criteria:

* Subjects with anatomical abnormalities of the genital tract.
* allergy to the drugs used for treatment.
* Y chromosome deletions or abnormal karyotypes.
* Subjects combined with cardiovascular, liver, kidney ,or hematopoietic system severe primary disease,or mental disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Sperm retrieval rate (SRR) | 4 months
  Semen analysis was performed every month from the end of the 6th month (two months after the last injection of hMG) to the end of 9th month until any sperm was found in the semen. If not sperm was found at the end of the 9th month, testicular sperm aspiration(TESA) was performed and the tissue was used for histological assessment. If any sperm was found in the semen analysis or TESA, the treatment was effective. The sperm retrieval rate was calculated.

SECONDARY OUTCOMES:
Hormonal profile | 9 months
  Serum FSH, LH, Total Testosterone, inhibin B were measured before the treatment and every month after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Yao, MD, Study Director — Center for Reproductive Medicine, Jinling Hospital, Medical School of Nanjing University
Locations (1):
- Center for Reproductive Medicine, Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hu X, Ding Z, Hong Z, Zou Z, Feng Y, Zhu R, Ma J, Ge X, Li C, Yao B. Spermatogenesis improved by suppressing the high level of endogenous gonadotropins in idiopathic non-obstructive azoospermia: a case control pilot study. Reprod Biol Endocrinol. 2018 Sep 22;16(1):91. doi: 10.1186/s12958-018-0401-7. PMID 30243299